CLINICAL TRIAL: NCT00443768
Title: Medication Review in Patients on Anti-parkinson Therapy
Acronym: PDCom
Status: Completed | Type: Observational
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Donald Grosset, Consultant Neurologist, South Glasgow University Hospitals NHS Trust
Other Study IDs: R060112/SW
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Parkinson's Disease
Keywords: Medication; Diagnosis; Community
MeSH Terms: conditions — Parkinson Disease; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
To identify patients within the community taking anti-parkinson medications in whom the diagnosis of Parkinson's disease is incorrect and to supervise and clinically monitor the withdrawal of anti-parkinson medications in this patient group

DETAILED DESCRIPTION:
Step 1 - Practice based pharmacist and medical review using database search for the following:

* Anti-parkinson drug therapy (excluding anticholinergic monotherapy).
* Disease codes to identify Parkinson's disease and parkinsonism, and exclude other diagnoses where anti-parkinson therapy may be used, although both are expected to be very small numbers (pituitary tumour, restless leg syndrome)
* To identify the duration of parkinsonism from the date of entry of the disease code.
* Pharmacy re-fill data to identify intermittent usage of treatment as an indicator of it being unlikely that the patient has idiopathic or dopa responsive parkinsonism.
* To identify patients on monotherapy with anti-parkinson therapy e.g. Selegiline for a prolonged duration as this is likely to suggest an alternative diagnosis.
* To record drug dosage over time, e.g. on an annual basis, again to identify whether patients fit in with the expected rates of change for degenerative parkinsonism where increasing combinations of drugs at higher doses are used over time.

Step 2 - Review of case records:

· Parkinson's disease nurse specialist and medical review of case records to identify additional clinical features of the condition and assist in identifying cases where it appears likely that anti-parkinson drug treatment is not helping the patient's condition.

Step 3 - Specialist out-patient review and follow-up:

· Invitation to the patient to attend the combined neurology/medicine for the elderly movement disorder clinic service where scoring against diagnostic clinical criteria would be undertaken, and where appropriate tapering of anti-parkinson therapy gradually under continued specialist observation.

ELIGIBILITY:
Inclusion Criteria:

Patients on anti-parkinson medication who:

* Have been on monotherapy for a prolonged period, or
* Use anti-parkinson medications intermittently, or
* Do not have the expected change in medication over time in keeping with degenerative Parkinson's disease.

Exclusion Criteria:

* Patients on anti-parkinson medication for reasons other than Parkinson's disease.
* Patients with significant co-morbidity (end stage liver, cardiac or renal disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample of Parkinson's disease patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Grosset, MD, Study Chair — Dept of Neurology, INS, Southern General Hospital; Edward Newman, MRCP, Principal Investigator — Dept of Neurology, INS, Southern General Hospital
Locations (1):
- Southern General Hospital, Glasgow, Scotland, United Kingdom